CLINICAL TRIAL: NCT04727567
Title: Effect of a Personalized Care Management Program on Hospital Inpatient Stays Among High Utilizers: A Randomized Clinical Trial
Brief Title: Evaluation of a Personalized Care Management Program for High Hospital Utilizers
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00082498; 04-20-10E (Other: Atrium)
Record Dates: First submitted 2021-01-12; First posted 2021-01-27 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-09

CONDITIONS: Comorbidities and Coexisting Conditions
Keywords: Patient Care Management; Patient Hospital Admissions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Visit Patient (MVP) Program: The MVP program aims to manage health and lower hospital utilization among patients with a history of high inpatient hospital stays at Atrium Health. Patients eligible for the program have four or more inpatient visits over the 12-month period prior to enrollment. Once enrolled, each MVP program participant receives on-going support from an assigned MVP care manager and larger care management team, including the following core program components:
  customized care plan developed for each patient at the time of enrollment routine, virtual health monitoring and collaborative care management team-based review personalized navigation and coordination across multidisciplinary Atrium Health services, as needed.
  Education, health coaching, and support via telephonic and in-person interactions, as needed.
- Usual Care: Atrium Health standard of care. Patient's post-discharge usual care depends on the inpatient care management assessment at last hospital admission. Patients can be discharged to home and receive no further care, or home with home health, or to a skilled nursing facility (SNF) or another type of Continuing Care facility. Patients can be referred to advanced illness management, hospice, and Community Care Partners by the inpatient care manager. Patient can be referred to Ambulatory Care Management for care management also via telehealth, by a primary care physician or the Transitions Clinic.

SUMMARY:
This randomized clinical trial intends to evaluate the effectiveness of enrollment in Atrium Health's Multiple Visit Patient (MVP) care management program compared to usual care on reducing 12-month total inpatient hospital utilization among patients with high past volume of hospital inpatient stays.

DETAILED DESCRIPTION:
The list of patients with four or more inpatient hospital visits in 2019 will be pulled from the Atrium Health electronic data warehouse (EDW) by IAS Clinical Quality Analytics, and eligibility for the MVP program of patients on this list will be determined by the Population Health's Care Management team based on predefined eligibility criteria. IAS CORE will randomize eligible participants into one of two groups: 1) MVP program; or 2) usual care.

Population Health's Multiple Visit Patient (MVP) care management program aims to manage health and lower hospital utilization among patients with a history of high inpatient hospital stays at Atrium Health. Patients eligible for the program have four or more inpatient visits over the 12-month period prior to enrollment. Once enrolled, each MVP program participant receives on-going support from an assigned MVP care manager and larger care management team, including the following core program components:

1. customized care plan developed for each patient at the time of enrollment
2. routine, virtual health monitoring and collaborative care management team-based review
3. personalized navigation and coordination across multidisciplinary Atrium Health services, as needed
4. education, health coaching, and support via telephonic and in-person interactions, as needed

The control group will receive usual care.

Upon completion of the 12-month period during which outcomes data will be accrued, the study will evaluate whether 12-month participation in the MVP program care management program, compared to usual care, reduced inpatient hospital use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* 4 or more inpatient hospital visits across Atrium Health Metro hospitals in 2019

Exclusion Criteria:

* Existing MVP participants
* Patients who at the time of identification for the MVP program are:
* Actively enrolled in a Levine Cancer Institute oncology navigation program
* Actively receiving hospice or palliative care
* Attributed to a primary care provider at an outside healthcare system
* Patients whose primary residence is a skilled nursing facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the evaluable population for this project, will have their data inform the final outcomes assessment. All patients who meet the inclusion and exclusion criteria in both groups will be assessed for the primary outcome (intent to treat).
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Number of inpatient (IP) hospital encounters over a 12 month period | 12 months
  Inpatient encounter is defined as an admission to an Atrium Health acute care hospital

SECONDARY OUTCOMES:
Number of inpatient hospital encounters over a 6 month period | 6 months
  Inpatient encounter is defined as an admission to an Atrium Health acute care hospital
Combined Inpatient and Observational hospital encounters - Atrium only | 6 months
  Combined number of IP and OBS encounters at Atrium Health hospitals
Combined Inpatient and Observational hospital encounters - non-Atrium included | 6 months
  Combined number of IP and OBS encounters at Atrium Health and non-Atrium Health hospitals
Combined Inpatient and Observational hospital encounters - Atrium only | 12 month
  Combined number of IP and OBS encounters at Atrium Health hospitals
Combined Inpatient and Observational hospital encounters - non-Atrium included | 12 month
  Combined number of IP and OBS encounters at Atrium Health and non-Atrium Health hospitals
Inpatient Readmission | 6 month
  Among patients with at least 1 encounter during the study period, 30-day all cause non-elective inpatient readmission rate to any AH hospital
Inpatient Readmission | 12 month
  Among patients with at least 1 encounter during the study period, 30-day all cause non-elective inpatient readmission rate to any AH hospital
Inpatient Readmission - Same Hospital | 6 month
  Among patients with at least 1 encounter during the study period, 30-day all cause non-elective inpatient readmission rate to the same AH hospital as the index encounter
Inpatient Readmission - Same Hospital | 12 month
  Among patients with at least 1 encounter during the study period, 30-day all cause non-elective inpatient readmission rate to the same AH hospital as the index encounter
Emergency Department Encounters | 6 month
  Number of patient emergency department encounters
Emergency Department Encounters | 12 month
  Number of patient emergency department encounters
Mortality | 6 month
  Dichotomous indicator of all-cause mortality within 6 months from the beginning of the study period
Mortality | 12 month
  Dichotomous indicator of all-cause mortality within 12 months from the beginning of the study period
Hospital Bed Days (Inpatient) | 6 month
  Total length of stay (LOS) in days (discharge date to admissions date) for acute care IP utilization
Hospital Bed Days (Inpatient) | 12 month
  Total length of stay (LOS) in days (discharge date to admissions date) for acute care IP utilization
Hospital Charges | 6 month
  Total accrued hospital billed charges for inpatient encounter at Atrium Health primary enterprise acute care facilities.
Hospital Charges | 12 month
  Total accrued hospital billed charges for inpatient encounter at Atrium Health primary enterprise acute care facilities.

CONTACTS AND LOCATIONS:
Overall Officials: Alica Sparling, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health - Care Management Program, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT04727567/Prot_SAP_000.pdf